CLINICAL TRIAL: NCT00579137
Title: CD45 and Alemtuzumab Monoclonal Antibody Conditioning Regimen For Allogeneic Donor Stem Cell Transplantation Of Patients With Severe Combined Immunodeficiency Disease (SCID) And Other Primary Immunodeficiency Disorders
Brief Title: Allogeneic SCT Of Pts With SCID And Other Primary Immunodeficiency Disorders
Acronym: MASCI
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Robert Krance, Professor Pediatrics Hematology Oncology Center for Cell and Gene Therapy, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21123-MASCI; NCT00609258 (obsolete NCT alias)
Record Dates: First submitted 2007-12-19; First posted 2007-12-21 (Estimated); Results first posted 2013-07-02 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Severe Combined Immunodeficiency Disease; Severe Primary Immunodeficiency Disorder; Undefined T Cell Deficiency Disorder; Wiskott-Aldrick Syndrome
Keywords: Severe Combined Immunodeficiency Disease; Severe Primary Immunodeficiency Disorder; Undefined T cell Deficiency Disorder; Wiskott-Aldrick Syndrome; Allogeneic stem cell transplant; Fludarabine; monoclonal antibodies
MeSH Terms: conditions — X-Linked Combined Immunodeficiency Diseases; Primary Immunodeficiency Diseases | interventions — Alemtuzumab; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Participants With SCID or Primary Immunodeficiency Disorder (Experimental): all patient will receive an allogeneic transplant with the following conditioning regimen Campath -1H, Fludarabine, Anti-CD45
  Interventions: Biological: Campath -1H; Drug: Fludarabine; Biological: Anti-CD45; Procedure: Stem cell infusion

INTERVENTIONS:
Biological: Campath -1H — Given intravenous on Days -8,-7, and -6
  Campath dose is weight based: for patients less than 15 kg the dose is 3 mg; for patients >15 kg to 30 kg the dose 5 mg; for patients > 30 kg the dose is 10 mg
  Other Names: Alemtuzumab
Drug: Fludarabine — Given intravenous on Days -8,-7,-6,-5, and -4
  Dose is 30 mg/m2
  Other Names: Fludara
Biological: Anti-CD45 — Given intravenous over 6 hours on Days -5,-4,-3, and -2
  Dose is 400 microgram/kg
Procedure: Stem cell infusion — stem cells are infused on day 0

SUMMARY:
This study is to discover whether children with severe combined immunodeficiency disease (SCID) or other primary immunodeficiency disorder (PID) for which no satisfactory treatment other than stem cell transplantation (SCT) exists can be safely and effectively transplanted from HLA mismatched (up to one haplotype) related donors or unrelated matched or mismatched (up to one antigen) donors, when leukocytolytic monoclonal antibodies (MAb) and Fludarabine are the sole conditioning agents. Three monoclonal antibodies will be used in combination. Two of them are rat IgG1 (immunoglobulin G1) antibodies directed against two contiguous epitopes on the CD45 (common leucocyte) antigen. They have been safely administered as part of the conditioning regimen for 12 patients receiving allografts (HLA matched and mismatched) at this center. They produce a transient depletion of >90% circulating leucocytes. The third MAb is Campath 1H, a humanized rat anti-CD52 MAb. Campath 1H, Alemtuzumab, has been licensed to treat B-cell chronic lymphocytic leukemia (B-CLL) and more recently has been safely given at this and other centers as part of a sub-ablative conditioning regimen to patients with malignant disease. Because these MAb produce both profound immunosuppression and significant, though transient, myelodestruction we believe they may be useful as the sole conditioning regimen in patients with SCID, in whom the use of conventional chemotherapeutic agents for conditioning may produce or aggravate unacceptable and even lethal short term toxicity. We anticipate MAb mediated subablative conditioning will permit engraftment in a high percentage of these patients with little or no immediate or long term toxicity. Campath IH persists in vivo for several days after administration and so will be present over the transplant period to deplete donor T cells as partial GvHD prophylaxis. Additional Graft versus Host Disease (GvHD) prophylaxis may be provided by administration of FK506.

DETAILED DESCRIPTION:
Donor Stem Cell Processing for Mismatched Donors: Harvested peripheral blood stem cells will be enriched for CD34 cells using the CliniMACS CD34 Reagent system, according to Center for Cell and Gene Therapy (CAGT) SOPs.

Stem Cell Transplant Conditioning

Campath-1H will be given as 3 daily intravenous infusions and will be followed by Anti-CD45 which will be given as four daily intravenous infusions that will be completed two days prior to stem cell infusion. Diphenydramine will be administered i.v. q4h during the period of the course of the Campath and Anti-CD45 infusions.

Day

8 Campath 1H as per CAGT SOP Fludarabine 10 kg or less: 1 mg/kg; > 10 kg: 30 mg/m2

7 Campath 1H as per CAGT SOP Fludarabine 10 kg or less: 1 mg/kg; > 10 kg: 30 mg/m2

6 Campath 1H as per CAGT SOP Fludarabine 10 kg or less: 1 mg/kg; > 10 kg: 30 mg/m2

5 YTH 24/54 400ug/kg over 6 hr Fludarabine 10 kg or less: 1 mg/kg; > 10 kg: 30 mg/m2

4 YTH 24/54 400ug/kg over 6 hr Fludarabine 10 kg or less: 1 mg/kg; > 10 kg: 30 mg/m2

3 YTH 24/54 400ug/kg over 6 hr

2 YTH 24/54 400ug/kg over 6 hr

1 rest

0 Stem Cell Infusion

Campath 1H Infusion- Campath dose is weight based: for patients less than 15 killograms (kg) administer Campath 3 mg; for patients >15 kg to 30 kg administer Campath 5 mg; for patients > 30 kg administer Campath 10 mg. Campath will be dosed and administered as per CAGT SOP.

Anti-CD45- Infusion Anti-CD45 infusion will be administered according to CAGT SOPs. 3 ml of heparinized blood will be drawn 48 hr post Anti-CD45 to evaluate for free Anti-CD45 levels in the plasma. This estimation will be used to determine whether treatment with irradiated leukocytes is required before the bone marrow is infused.

GVHD Prophylaxis- GVHD prophylaxis will be achieved through positive selection for CD34 resulting in > 3 log T cell depletion. Previous reports have indicated that there is a low frequency of severe (Grade II/IV) GVHD after haploidentical transplants if recipients receive stem cell populations containing <5 x 10 CD3 positive T cells. We hope to achieve such levels with our CD34 enrichment protocol. However, pharmacologic prophylaxis will be added if the CD34 selected product contains more than 5 x 10 CD3+ve T cells/kg recipient weight. In addition, Campath 1H persists in the recipient circulation through the immediate transplant period and will contribute anti-GVHD activity, in vivo. Patients who develop acute or chronic GVHD will be managed according to CAGT SOPs.

ELIGIBILITY:
Inclusion Criteria:

- Patients with a diagnosis of: Severe combined immunodeficiency disease

This includes patients whose SCID is characterized by gene specific mutations as well as patients with clinically severe combined immunodeficiency without a defined genetic cause in which the diagnosis will be determined by a combination of clinical course with lymphocyte quantification and function assays.

OR

Severe primary immunodeficiency disorder, including undefined T cell deficiency disorder, Wiskott-Aldrich syndrome, and other severe immunodeficiencies for which satisfactory conventional therapy does not exist.

* Availability of an HLA mismatched (up to one haplotype) family member or an HLA matched or mismatched (up to one antigen) unrelated donor.
* Creatinine < 2.5 x normal for age.
* Life expectancy greater than 6 weeks
* Lansky/Karnofsky greater than or equal to 70%

Exclusion Criteria:

* Patients with an HLA matched related donor
* Patients with symptomatic cardiac disease, or evidence of significant cardiac disease by echocardiogram (i.e., shortening fraction less than 25%)
* Patients with known allergy to rat serum products
* Patients with a severe infection that on evaluation by the Principal Investigator precludes ablative chemotherapy or successful transplantation
* HIV positive
* Pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Krance, MD, Principal Investigator — Baylor College of Medicine; Malcolm Brenner, MD, Study Chair — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With SCID or Primary Immunodeficiency Disorder: Participants received an allogeneic stem cell transplant with the following conditioning:
  Day 8 Campath 1H as per CAGT SOP, Fludarabine 10 kg or less: 1 mg/kg; > 10 kg: 30 mg/m2
  D7 Campath 1H as per CAGT SOP, Fludarabine 10 kg or less: 1 mg/kg; > 10 kg: 30 mg/m2
  D6 Campath 1H as per CAGT SOP, Fludarabine 10 kg or less: 1 mg/kg; > 10 kg: 30 mg/m2
  D5 Anti-CD45 MAb 400ug/kg over 6 hr, Fludarabine 10 kg or less: 1 mg/kg; > 10 kg: 30 mg/m2
  D4 Anti-CD45 MAb 400ug/kg over 6 hr, Fludarabine 10 kg or less: 1 mg/kg; > 10 kg: 30 mg/m2
  D3 Anti-CD45 MAb 400ug/kg over 6 hr
  D2 Anti-CD45 MAb 400ug/kg over 6 hr
  D1 rest
  D0 Stem Cell Infusion
  Campath dose is weight based: for patients less than 15 kg administer Campath 3 mg; for patients >15 kg to 30 kg administer Campath 5 mg; for patients > 30 kg administer Campath 10 mg. Campath will be dosed and administered as per CAGT SOP.
  Anti-CD45 infusion will be administered according to CAGT SOPs.
Period: Overall Study
Arm/Group | Participants With SCID or Primary Immunodeficiency Disorder
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Group: only one group
Arm/Group | Single Group
Number analyzed (Participants) | 3
Age, Customized [Number; unit: participants]
  <=1 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Donor Engraftment
Time Frame: 100 Days
Measure: Number; unit: participants
Arm/Group | Single Group
Number analyzed (Participants) | 3
participants | 1

2. Secondary Outcome: Patients Alive at 1 Year
Time Frame: 1 Year
Measure: Number; unit: participants
Arm/Group | Single Group
Number analyzed (Participants) | 3
participants | 3

3. Secondary Outcome: Number of Patients With Grade III or IV Toxicity
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | Single Group
Number analyzed (Participants) | 3
participants | 0

4. Secondary Outcome: Number of Patients With Grade III to IV Acute GVHD
Time Frame: 100 days
Measure: Number; unit: participants
Arm/Group | Single Group
Number analyzed (Participants) | 3
participants | 0

ADVERSE EVENTS:
Arm/Group | Single Group
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Group (N=3)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 1 (5)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (5)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Dermatology/Skin - Other: Livedo reticularis (Skin and subcutaneous tissue disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (5)
Hepatobiliary/Pancreas - Other: Liver GvHD (Hepatobiliary disorders) | 1 (1)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils - Catheter-related (Infections and infestations) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (17)
Lymphopenia (Blood and lymphatic system disorders) | 1 (23)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (10)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 1 (1)
Pain - Abdomen NOS (General disorders) | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 1 (4)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (7)
Pulmonary/Upper Respiratory - Other: Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1 (3)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (5)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 1 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes